CLINICAL TRIAL: NCT05933798
Title: China Pilot of ICOPE (Integrated Care for Older People) in Chaoyang District, Beijing
Brief Title: China Pilot of ICOPE (Integrated Care for Older People) in Chaoyang
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pinetree Health Technologies (Beijing) Co., Ltd. (Industry)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-QS-001
Record Dates: First submitted 2023-06-06; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Aging; Healthy Aging; Utilization, Health Care
Keywords: integrated care; primary care; ICOPE; decade of healthy ageing
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants who were actively followed up during the study period with a personalized integrated care plan developed following the ICOPE screening and assessment, identified as "at-risk" for loss in intrinsic capacity.
  Interventions: Other: ICOPE
- Control Group (Active Comparator): Pariticpants who continued receiving usual care during the study period.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ICOPE — The ICOPE approach with locally adapted care pathways was implemented by trained integrated care managers (ICMs) advised by multi-disciplinary teams, delivered in primary care settings
  Arms: Intervention Group
Other: Usual Care — Participants in the Control Group would have their care plan after assessment and seek health and care services as usual without additional advice or support on implementing the care plan
  Arms: Control Group

SUMMARY:
The goal of this pilot study is to examine predefined parameters (sample size, capacity building, acceptance by community-dwelling older people (participants) and care providers) to evaluate the feasibility of implementing World Health Organization's ICOPE (integrated care for older people) approach in China. The main questions it aims to answer are:

1. Whether it is feasible to implement the ICOPE approach in China;
2. Whether the integrated care approach would make any difference in health outcomes and resource utilization.

Participating older adults receiving integrated care (Intervention Group) are compared to those receiving usual care (Control Group) in order to answer the two questions above.

DETAILED DESCRIPTION:
The goal of this pilot study is to evaluate the feasibility of implementing World Health Organization's ICOPE (integrated care for older people) approach in China. The main questions it aims to answer are:

1. Whether it is feasible to implement the ICOPE approach in China;
2. Whether the integrated care approach would make any difference in health outcomes and resource utilization.

For the first question, predefined parameters such as sample size, capacity building, acceptance by community-dwelling older people (participants) and care providers were examined.

Based on literature review and also as evidenced in the background study of the ICOPE guideline development process, a key hypothesis is that implementing integrated care management programs can improve health outcomes while containing costs.

According to the pilot study design, a total of 2000 community-dwelling older persons aged 60 and above at-risk of functional loss in Chaoyang District of Beijing are recruited and randomly assigned to the intervention group (n=500) and control group (n=1500).

Chaoyang is the most populated district in Beijing, with subdistricts that are urban, suburban and rural, well representing the city of Beijing. To identify potential participants who are at risk of functional loss, the pilot used ICOPE screening tools in the recruitment process, to screen for any losses in mobility, cognition, vitality, psychological health, vision and hearing.

Screening tools used are:

1. Independence is measured by the activities of daily living (ADL) 14-questionnaire scale.
2. Cognition is measured by mini-mental status examination (MMSE).
3. Vitality or nutrition is measured by by mini-nutritional assessment- short form (MNA-SF) to assess the risk of malnutrition.
4. Mobility is measured by short physical performance battery (SPPB).
5. Psychological health is measured by geriatric depression scale-five items (GDS-5).

ELIGIBILITY:
Inclusion Criteria:

* Screened as positive for intrinsic capacity declines
* Decline in intrinsic capacity confirmed by in-depth assessment in any of the domains described as: MMSE < 27 (for cognition), SPPB ≤ 9 (for locomotion), MNA-SF <12 (for vitality we used nutrition as a proxy), GDS-5 ≥ 2 (for psychology we used depression as a proxy) or any vision impairment
* Signed form of consent and willingly participate in the pilot study

Exclusion Criteria:

* Negative results in their intrinsic capacity decline screening
* Severe hearing problems as the study was conducted during COVID-19 pandemics period and relied on telecare or remote sessions of intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2148 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing the ICOPE program in China | 12 months
  1. Sample size (to successfully recruit over 2,000 participants, 500 of whom were to be categorized in the intervention group)
  2. Capacity building (at least 200 primary care providers to be fully trained and deployed in the pilot program)
  3. Acceptance (reach more than 90% satisfaction with the pilot by both participants and providers).

SECONDARY OUTCOMES:
Independence | 6 months
  measured by the activities of daily living (ADL) 14-questionnaire scale, to assess the participant's physical function
Cognition | 6 months
  measured by mini-mental status examination (MMSE) to assess the cognitive health of the participants
Vitality | 6 months
  nutrition measured by mini-nutritional assessment- short form (MNA-SF) to assess the risk of malnutrition
Mobility | 6 months
  measured by short physical performance battery (SPPB) to assess the risk of declining mobility
Psychological health | 6 months
  measured by geriatric depression scale-five items (GDS-5) using a short set of questions to assess possible depressive symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ninie Wang, MBA DrPH, Principal Investigator — Pinetree Care Group
Locations (1):
- Pinetree Care Group, Beijing, China

IPD SHARING:
Plan to Share IPD: No
Access to de-identified data of the China ICOPE Pilot (2020-2021) by other researchers is subject to the approval of an independent review committee and after signing a data access and a data use agreement.

REFERENCES:
- [Background] Tavassoli N, de Souto Barreto P, Berbon C, Mathieu C, de Kerimel J, Lafont C, Takeda C, Carrie I, Piau A, Jouffrey T, Andrieu S, Nourhashemi F, Beard JR, Soto Martin ME, Vellas B. Implementation of the WHO integrated care for older people (ICOPE) programme in clinical practice: a prospective study. Lancet Healthy Longev. 2022 Jun;3(6):e394-e404. doi: 10.1016/S2666-7568(22)00097-6. Epub 2022 Jun 9. PMID 36098317
- See also: WHO's report on findings from implementing ICOPE pilots in different countries — https://www.who.int/news/item/25-04-2022-integrated-care-for-older-people--who-launches-new-report-of-findings-from-the-icope-implementation-pilot-programme

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT05933798/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT05933798/ICF_001.pdf